CLINICAL TRIAL: NCT00066599
Title: An Open-Label, Intravenous To Oral Switch, Multiple Dose, Multi-Center Study To Investigate The Pharmacokinetics, Safety And Tolerability Of Voriconazole In Hospitalized Children Aged 2 - <12 Years Who Require Treatment For The Prevention Of Systemic Fungal Infection
Brief Title: Voriconazole in Preventing Fungal Infections in Children With Neutropenia After Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000316329; NCI-03-C-0218; NCT00062920 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-07

CONDITIONS: Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Neuroblastoma; Neutropenia; Sarcoma
Keywords: neutropenia; recurrent childhood lymphoblastic lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; recurrent/refractory childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; childhood acute promyelocytic leukemia (M3); previously treated childhood rhabdomyosarcoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood rhabdomyosarcoma; childhood chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; acute undifferentiated leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; secondary acute myeloid leukemia; untreated childhood acute lymphoblastic leukemia; disseminated neuroblastoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent neuroblastoma; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Neutropenia; Sarcoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Recurrence; Wilms Tumor; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Voriconazole

INTERVENTIONS:
Drug: voriconazole

SUMMARY:
RATIONALE: Voriconazole may be effective in preventing systemic fungal infections following chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of voriconazole in preventing systemic fungal infections in children who have neutropenia after receiving chemotherapy for leukemia, lymphoma, or aplastic anemia or in preparation for bone marrow or stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetics of voriconazole administered IV and orally for the prevention of systemic fungal infection in pediatric patients with neutropenia after chemotherapy.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is a pilot, open-label, multicenter study. Patients are stratified according to age (2 to 5 vs 6 to 11).

Within 48 hours after completion of chemotherapy, patients begin prophylactic therapy:

* Cohort 1 (the first 18 patients, 9 per stratum): Patients receive voriconazole IV over 80-160 minutes twice daily on days 1-8 and oral voriconazole* twice daily beginning on day 9.

Depending on the results of the interim pharmacokinetic analysis, the last 18 patients entered on the study receive 1 of the following regimens:

* Cohort 2A:Patients receive voriconazole as in cohort 1 at a higher dose.
* Cohort 2B: Patients receive voriconazole IV over 80-160 minutes twice daily on days 1-4 and oral voriconazole* twice daily beginning on day 5.

NOTE: *Patients who are unable to tolerate oral medication may continue receiving IV medication until day 20.

In all cohorts, treatment continues until blood counts recover or day 30 in the absence of unacceptable toxicity or progression of infection.

Patients are followed at 30 days and at 12 months.

PROJECTED ACCRUAL: A total of 49 patients (approximately 24 per stratum) were accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Expected to develop neutropenia (absolute neutrophil count less than 500/mm^3) lasting for more than 10 days after chemotherapy for 1 of the following conditions:

  * Leukemia
  * Lymphoma
  * Aplastic anemia
  * Preparation for a bone marrow or stem cell transplantation
* Requiring treatment for the prevention of systemic fungal infection

PATIENT CHARACTERISTICS:

Age

* 2 to 11

Performance status

* Not specified

Life expectancy

* More than 3 months

Hematopoietic

* See Disease Characteristics

Hepatic

* AST and ALT no greater than 5 times upper limit of normal (ULN)
* Bilirubin no greater than 5 times ULN

Renal

* Creatinine clearance at least 30 mL/min

Cardiovascular

* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* No severe hypokalemia (potassium less than 3.2 mmol/L)
* No prior hypersensitivity to or severe intolerance of azole antifungal agents
* No other concurrent condition that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 24 hours since prior use of any of the following:

  * Terfenadine
  * Pimozide
  * Quinidine
  * Astemizole
  * Cisapride
  * Omeprazole
* More than 14 days since prior use of any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenytoin
  * Nevirapine
  * Long-acting barbiturates
* No prior sirolimus
* No prior enrollment on this study
* No concurrent use of any of the following:

  * Terfenadine
  * Pimozide
  * Quinidine
  * Astemizole
  * Cisapride
  * Omeprazole
* No other concurrent investigational drugs except any of the following:

  * Drugs used as treatment for cancer
  * Antiretroviral agents
  * Drugs used for the treatment of any AIDS-defining opportunistic infections
* No concurrent enrollment in investigational anticancer drug trials that exclude the use of other investigational agents

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-06; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (7):
- United States (7):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital and Health Center, San Diego, San Diego, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas